CLINICAL TRIAL: NCT04779606
Title: A Phase I/II, Randomized, Placebo-controlled, Double-masked, Efficacy, Safety and Local Tolerability Study of Chloroprocaine 3% Gel Eye Drops in Healthy Volunteers
Brief Title: Efficacy, Safety and Local Tolerability Study of Chloroprocaine 3% Gel Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHL.3-01-2020
Record Dates: First submitted 2021-01-19; First posted 2021-03-03 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine (Experimental): Chloroprocaine 3% ocular gel (30 mg/mL), 3 drops instilled at a 1 min ± 15 sec interval.
  Interventions: Drug: Ocular gel
- Placebo (Placebo Comparator): Vehicle for chloroprocaine 3% ocular gel, 3 drops instilled at a 1 min ± 15 sec interval.
  Interventions: Drug: Ocular gel

INTERVENTIONS:
Drug: Ocular gel — 3 drops instilled in the right eye
  Other Names: No other intervention names

SUMMARY:
The study evaluate the efficacy, safety and local tolerability of Chloroprocaine 3% ophthalmic gel as compared to matching placebo in healthy subjects.

DETAILED DESCRIPTION:
One hundred and five (105) healthy male and female subjects will be randomised in a 4:1 ratio to receive a single ocular instillation of Chloroprocaine 3% ophthalmic gel or matching placebo (vehicle) (84 subjects will receive chloroprocaine and 21 subjects will receive placebo). The assigned investigational product (3 drops) will be instilled in the right eye of each subject. Administrations will be performed at the clinical centre by the Investigator or his deputy on study day 1. For each administration, the 3 drops will be instilled at a 1 min ± 15 sec interval.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Signed written informed consent before inclusion in the study
* Sex and age: Healthy men and women, 18 - 55 years inclusive
* Body Mass Index: 18.5-30 kg/m2 inclusive
* Vital signs: Systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Contraception and fertility: women of child-bearing potential must be using at least one of the following reliable methods of contraception:

  1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit;
  2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
  3. A male sexual partner who agrees to use a male condom with spermicide
  4. A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all women, urine pregnancy test result must be negative at screening.

Exclusion Criteria:

* Physical findings: Clinically significant abnormal physical findings which could interfere with the objectives of the study
* Visual acuity: Best corrected visual acuity < 1/10
* Concomitant medications: Medications, including over the counter medications and herbal remedies, systemic opioids and morphine drugs, topical ocular products with anaesthetic action, systemic analgesic drugs, for 2 weeks before study screening
* Ophthalmic diseases: Clinically significant ocular disease; eye movement disorder (i.e. nystagmus); dacryocystitis and all others pathologies of tears drainage system; corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration and superficial punctuate keratitis); history of inflammatory ocular disease (iritis, uveitis, herpetic keratitis), history of ocular traumatism, infection or inflammation within the last 3 months or history of any other ocular disease that may affect the outcome of the study or the subject's safety
* Ophthalmic surgery: History of ophthalmic surgical complications (e.g. cystoid macular oedema) in the last 6 months
* Diseases: Significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, psychiatric or neurological diseases or surgeries that may interfere with the aim of the study
* Allergy: Ascertained or presumptive hypersensitivity to the active principle and/or ingredients of investigational products; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol [greater than 1 drink/day for women and greater than 2 drinks/day for men, defined according to the USDA Dietary Guidelines 2015-2020], caffeine (greater than 5 cups coffee/tea/day) or tobacco abuse (greater than or equal 10 cigarettes/day)
* Alcohol test: positive alcohol breath test at Day 1
* Pregnancy (women only): positive or missing pregnancy test at screening, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, Principal Investigator — CROSS Research S.A., Phase I Clinical Unit, Arzo, Switzerland
Locations (1):
- CROSS Research S.A., Arzo, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: First Phase: Tolerability and Safety
Arm/Group | Chloroprocaine | Placebo
Started | 16 | 4
Completed | 16 | 4
Not Completed | 0 | 0
Period: Second Phase: Efficacy
Arm/Group | Chloroprocaine | Placebo
Started | 68 | 17
Completed | 68 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Placebo | Total
Number analyzed (Participants) | 84 | 21 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.8) | 37.3 (10.9) | 38.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 10 | 62
  Male | 32 | 11 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 79 | 20 | 99
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 84 | 21 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Gaining Full Conjunctival Anesthesia of the Ocular Surface
Description: Number of partecipants gaining full conjunctival anesthesia of the ocular surface, evaluated by conjunctiva pinching (0.3-mm forceps), 5 minutes after administration of Chloroprocaine 3% ophthalmic gel, in comparison to placebo - only study eye (right eye)
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 68 | 17
Participants | 61 | 2

2. Secondary Outcome: Time to Anesthesia, Evaluated by Conjunctiva Pinching (0.3-mm Forceps) - Only Study Eye (Right Eye)
Description: Time to anesthesia, evaluated by conjunctiva pinching (0.3-mm forceps) - only study eye (right eye)
Time Frame: Day 1
Population: A total of 105 healthy men and women were planned and enrolled included in the study. Initially, local tolerability and safety was evaluated in the first 20 enrolled subjects . After the first 20 subjects had completed the study, local tolerability and safety data were evaluated and treatment safety was confirmed according to the clinical study protocol specifications. Efficacy, beside local tolerability and safety, was assessed in the 85 subsequent subjects
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 68 | 17
minutes | 2.41 (2.12) | 4.49 (1.44)

3. Secondary Outcome: Duration of Anesthesia - Only Right Eye
Description: Duration of anesthesia, evaluated by conjunctiva pinching (0.3-mm forceps) - only study eye (right eye)
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 68 | 17
minutes | 18.3 (10) | 19.3 (14)

4. Secondary Outcome: Visual Acuity (EDTRS Chart) - Both Eyes
Description: Visual acuity will be assessed, for all subjects and both eyes using an EDTRS chart (visual acuity is scored with reference to the logarithm of the minimum angle of resolution, an observer who can resolve details as small as 1 minute of visual angle scores LogMAR 0, since the base-10 logarithm of 1 is 0; an observer who can resolve details as small as 2 minutes of visual angle (i.e., reduced acuity) scores LogMAR 0.3, since the base-10 logarithm of 2 is near-approximately 0.3; and so on)
Time Frame: Up to day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 68 | 17
LogMAR
  screening right eye | 1 (0.1) | 0.9 (0.2)
  follow up right eye | 1 (0.1) | 1 (0.1)
  screening left eye | 1 (0.2) | 1 (0.1)
  follow up left eye | 1 (0.1) | 1 (0.1)

5. Secondary Outcome: Ocular Symptoms
Description: The ocular symptoms will be assessed: burning, stinging, itching, foreign body sensation.
  Scores will be determined using a 100 mm VAS where 0 means "no symptoms" and 100 means "worst possible discomfort".
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
mm
  burning in right eye at Screening | 0 (0) | 0 (0)
  burning in right eye at pre-dose | 0 (0) | 0 (0)
  burning in right eye at post-dose | 1.17 (10) | 0.14 (0.65)
  burning in right eye at follow-up | 1.35 (10.8) | 0 (0)
  Stinging in right eye at screening | 0 (0) | 0 (0)
  Stinging in right eye at pre-dose | 0 (0) | 0 (0)
  Stinging in right eye at post-dose | 0.73 (6.66) | 0.05 (0.22)
  Stinging in right eye at follow-up | 1.88 (12.51) | 0 (0)
  Itching in right eye at screening | 0 (0) | 0 (0)
  Itching in right eye at pre-dose | 0 (0) | 0 (0)
  Itching in right eye at post-dose | 1.17 (10.05) | 0.14 (0.65)
  Itching in right eye at follow-up | 1.35 (10.8) | 0 (0)
  Foreign body sensation in right eye at screening | 0 (0) | 0 (0)
  Foreign body sensation in right eye at pre-dose | 0 (0) | 0 (0)
  Foreign body sensation in right eye at post-dose | 0.93 (6.12) | 0.33 (1.06)
  Foreign body sensation in right eye at follow-up | 1.21 (7.92) | 0 (0)

6. Secondary Outcome: Ocular Signs by Slit Lamp Examination
Description: Slit lamp biomicroscopy will be performed for the assessment of the following parameters:
  conjunctival redness, anterior chamber flare, conjunctival chemosis, eyelid swelling.
  Presence and severity will be graded according to a 4 point scale, where (0) none, (1) mild, (2) moderate, (3) severe.
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
score on a scale
  Conjunctival redness scores at screening | 0.04 (0.19) | 0.05 (0.22)
  Conjunctival redness scores at pre-dose | 0.02 (0.15) | 0 (0)
  Conjunctival redness scores at post dose | 0.29 (0.57) | 0.14 (0.48)
  Conjunctival redness scores at follow-up | 0 (0) | 0 (0)
  Anterior chamber flare at screening | 0 (0) | 0 (0)
  Anterior chamber flare at pre-dose | 0 (0) | 0 (0)
  Anterior chamber flare post-dose | 0 (0) | 0 (0)
  Anterior chamber flare follow-up | 0 (0) | 0 (0)
  Conjunctival chemosis at screening | 0 (0) | 0 (0)
  Conjunctival chemosis at pre-dose | 0 (0) | 0 (0)
  Conjunctival chemosis at post-dose | 0 (0) | 0 (0)
  Conjunctival chemosis at follow-up | 0 (0) | 0 (0)
  Eyelid swelling at screening | 0 (0) | 0 (0)
  Eyelid swelling at pre-dose | 0 (0) | 0 (0)
  Eyelid swelling post-dose | 0 (0) | 0 (0)
  Eyelid swelling at follow-up | 0 (0) | 0 (0)

7. Secondary Outcome: Corneal Fluorescein Staining by Slit Lamp Examination - Both Eyes
Description: Fluorescein will be used to detect corneal epithelial defects using slit lamp biomicroscopy. As grading scale for corneal damage, the NEI/Industry Workshop guidelines will be used. The cornea will be divided into five sectors (central, superior, inferior, nasal and temporal), each of which is scored on a scale of 0-3, where 0 means no staining and 3 means maximum staining, with a maximal score of 15.
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
score on a scale
  Screening - right eye | 0 (0.1) | 0 (0)
  follow-up - right eye | 0 (0.2) | 0 (0.2)
  screening - left eye | 0 (0.2) | 0 (0)
  follow-up - left eye | 0 (0.1) | 0 (0.2)

8. Secondary Outcome: Intraocular Pressure (IOP) - Both Eyes
Description: Intraocular pressure will be measured with a slit-lamp mounted Goldmann applanation tonometer. Before each measurement one drop of oxybuprocaine hydrochloride combined with sodium fluorescein will be used for local anaesthesia of the cornea.
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
mm Hg
  right eye at screening | 12.7 (2.6) | 13.2 (2.5)
  right eye at follow-up | 12.3 (2.1) | 12.3 (2.0)
  left eye at screening | 12.5 (2.3) | 13.5 (2.2)
  left eye at follow-up | 12.4 (2.2) | 12.6 (2.0)

9. Secondary Outcome: Fundus Ophthalmoscopy (Vitreous, Macula, Retina and Optic Nerve Head) With the Slit Lamp - Both Eyes
Description: Indirect fundus ophthalmoscopy will be performed, for all subjects and both eyes, with the observation at the slit lamp using a +90 diopters Volk lens.The evaluation is performed with a grading scale: 0 None, 1 Mild, 2 Moderate, 3 Severe for each parameters evaluated.
Time Frame: Up to day 7
Population: Initially, safety and local tolerability were evaluated and confirmed in the first 20 enrolled subjects. Then efficacy, beside local tolerability and safety, was assessed in the 85 additional subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
score on a scale
  Vitreous scores in right eye at screening | 0 (0) | 0 (0)
  Vitreous scores in right eye at follow up | 0 (0) | 0 (0)
  Vitreous scores in left eye at screening | 0 (0) | 0 (0)
  Vitreous scores in left eye at follow up | 0 (0) | 0 (0)
  Macula, (Peripheral) Retina and Optic Nerve scores in right eye at screening | 0 (0) | 0 (0)
  Macula, (Peripheral) Retina and Optic Nerve scores in right eye at follow up | 0 (0) | 0 (0)
  Macula, (Peripheral) Retina and Optic Nerve scores in left eye at screening | 0 (0.1) | 0 (0)
  Macula, (Peripheral) Retina and Optic Nerve scores in left eye at follow-up | 0 (0.1) | 0 (0)

10. Secondary Outcome: Vital Signs (Blood Pressure)
Description: Subjects blood pressure will be measured by the Investigator or his/her deputy
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
mmHg
  Systolic - predose | 115.6 (10.2) | 120.4 (10.4)
  systolic - postdose | 116 (11.8) | 115.3 (10.1)
  diastolic - predose | 71.7 (11.5) | 73.5 (10.1)
  diastolic - postdose | 72.0 (11.5) | 71 (10.6)

11. Secondary Outcome: Vital Signs (Heart Rate)
Description: Subjects heart rate will be measured by the Investigator or his/her deputy
Time Frame: Up to day 7
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Chloroprocaine | Placebo
Number analyzed (Participants) | 84 | 21
beats/minute
  pre-dose | 72.7 (10.1) | 70.7 (10)
  post-dose | 68.4 (8.8) | 67.3 (8.6)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Chloroprocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/21
Other Adverse Events (participants affected / at risk) | 27/84 | 4/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine (N=84) | Placebo (N=21)
Mydriasis (Eye disorders) | 16 (16) | 0 (0)
conjunctival Hyperemia (Eye disorders) | 10 (10) | 2 (2)
puncatte keratitis (Eye disorders) | 6 (6) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 5 (5) | 0 (0)
eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 2 (2)
eye irritation (Eye disorders) | 1 (1) | 0 (0)
eye pain (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT04779606/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT04779606/SAP_001.pdf